CLINICAL TRIAL: NCT06191822
Title: Aspire2B Personalization Pilot Study Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PEP- 2111/19 - 2302/07/08/09
Record Dates: First submitted 2023-09-13; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: App Proficiency; Behavior; Lifestyle
Keywords: Biological age; Wellness app
MeSH Terms: conditions — Behavior | interventions — Nutritional Status; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrition (Other): Set personalized nutrition goals
  Interventions: Other: Nutrition
- Fitness (Other): Set personalized fitness goals
  Interventions: Other: Fitness
- Sleep (Other): Set personalized sleep goals
  Interventions: Other: Sleep

INTERVENTIONS:
Other: Nutrition — Interact with mobile app and work toward personalized nutrition goals
  Arms: Nutrition
Other: Fitness — Interact with mobile app and work toward personalized fitness goals
  Arms: Fitness
Other: Sleep — Interact with mobile app and work toward personalized sleep goals
  Arms: Sleep

SUMMARY:
This non-randomized pilot study program is focused on assessing the technical characteristics of the Aspire2B mobile device application.

DETAILED DESCRIPTION:
Aspire2B is a mobile wellness app that uses non-invasive measurements to predict various physiological states and estimate biological age. Users are then enrolled in nutrition, fitness, or sleep challenges within the app that are aimed at improving overall wellness and thus helping to reduce biological age. Mobile health (mHealth) interventions require numerous decisions that integrate behavioral theory, user feedback, and technical and practical feasibility considerations. The main purpose of this research program is to test if the application works as intended. This pilot study program is managed internally by Pepsico clinical researchers.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in reading and understanding English or Spanish
* Smartphone users

Exclusion Criteria:

* Cannot proceed to onboarding without downloading the app, consenting to participate, and agreeing to app Terms of Use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess the technical characteristics of the app (App proficiency) -Connection | Continuous for up to 6 weeks
  Does the app work as intended: Ability to connect wearable devices
Assess the technical characteristics of the app (App proficiency) -Face scan age | Continuous for up to 6 weeks
  Does the app work as intended: Ability to conduct face scan to provide biological age
Assess the technical characteristics of the app (App proficiency) -Face scan stress | Continuous for up to 6 weeks
  Does the app work as intended: Ability to conduct face scan to provide stress index
Assess the technical characteristics of the app (App proficiency) -Face scan heart rate | Continuous for up to 6 weeks
  Does the app work as intended: Ability to conduct face scan to provide heart rate
Assess the technical characteristics of the app (App proficiency) -Onboarding | Continuous for up to 6 weeks
  Does the app work as intended: Onboarding sequence
Assess the technical characteristics of the app (App proficiency) -Goal selection | Continuous for up to 6 weeks
  Does the app work as intended: Ability to enter own goal
Assess the technical characteristics of the app (App proficiency) -Goal progress | Continuous for up to 6 weeks
  Does the app work as intended: Ability to track and measure goal progress (e.g., steps from a wearable device)
Assess the technical characteristics of the app (App proficiency) -Points assigned | Continuous for up to 6 weeks
  Does the app work as intended: Do points earned reflect what was completed in the app?
Assess the technical characteristics of the app (App proficiency) -Wellness scoring | Continuous for up to 6 weeks
  Does the app work as intended: Does wellness score change with lifestyle changes as intended?

SECONDARY OUTCOMES:
Learnings to inform future versions of the app -Retention | Continuous for up to 6 weeks
  Exploratory analyses of the data aimed to help to inform clinical trial retention rates
Learnings to Inform future versions of the app -Overall engagement | Continuous for up to 6 weeks
  Exploratory analyses of the data aimed to help to inform predictors of engagement
Learnings to inform changes to future versions of the app -Specific engagement | Continuous for up to 6 weeks
  Exploratory analyses of the data aimed at informing engagement with specific app features
Learnings to inform changes to future versions of the app - Dietary behaviors | Continuous for up to 6 weeks
  Exploratory analyses of the data aimed at informing improvements in self-reported diet behaviors
Learnings to inform changes to future versions of the app -Lifestyle behaviors | Continuous for up to 6 weeks
  Exploratory analyses of the data aimed at informing improvements in self-reported lifestyle behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Tristin Brisbois, PhD, MBS, Principal Investigator — PepsiCo Global R&D
Locations (1):
- Remote, no facility visits. Managed by PepsiCo R&D Life Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No